CLINICAL TRIAL: NCT02732912
Title: SleepSure: A Randomised Controlled Trial to Assess the Effects of Eye Masks and Earplugs on Hospital Inpatient Sleep
Brief Title: SleepSure: A Trial to Assess the Effects of Eye Masks and Earplugs on Hospital Inpatient Sleep
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Adam Monk, Principle Investigator, Oxford University Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SleepSure
Record Dates: First submitted 2016-03-31; First posted 2016-04-11 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Sleep
Keywords: falls; sleep
MeSH Terms: interventions — Ear Protective Devices; zopiclone

STUDY DESIGN:
Intervention Model Description: Randomised, investigator-blinded, parallel group design
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Patients in this arm will continue current standard management for sleep, which is largely reactive; if a patient requests night sedation or complains that they cannot sleep and that they want help, then zopiclone is prescribed, starting at 3.75 mg.
  Interventions: Drug: Zopiclone
- Eye mask and ear plugs (Experimental): General management will be as for the control group. In addition, patients in this group will be given ear plugs and eye shades (masks) to use when trying to sleep. The patient will generally be responsible for using or not using the equipment, though ward nurses may remind patients if they notice that the patient has the equipment.
  Interventions: Device: Ear plugs; Device: Eye Mask; Drug: Zopiclone

INTERVENTIONS:
Device: Ear plugs — The patient will be given a plastic wallet containing an eye mask and ear plugs, to be used when trying to sleep.
  Arms: Eye mask and ear plugs
Device: Eye Mask — The patient will be given a plastic wallet containing an eye mask and ear plugs, to be used when trying to sleep.
  Arms: Eye mask and ear plugs
Drug: Zopiclone — This night sedation will be given to any patient requesting it, in either group
  Other Names: Zimovane

SUMMARY:
The aim of this study is to determine whether routinely providing patients admitted to hospital with two devices to help sleep - ear plugs, and an eyeshade - leads to patients having a better quality of sleep and/or longer, more satisfying sleep.

DETAILED DESCRIPTION:
This is a prospective, investigator blinded, randomised controlled study involving all patients admitted to any of ten acute wards in a large, busy hospital serving both the local population of about 700,000 people and a wider area for specialist services.

Patients will be identified at the time of admission and recruited as soon as possible by nursing and medical staff involved in the admission process. The primary exclusion criterion is some obvious reason that using the equipment is not possible (e.g. allergy to materials used).

After gaining consent, from the patient, or assent from a relative if the person is unable to consent at the time, the patient will be registered and allocated a number. Each ward will have prefilled envelopes with a randomly determined group allocation within it, and after registration this will be opened to determine the patient's group. Each patient will be given a short information leaflet and consent form.

Patients allocated to the intervention will be given the ear plugs and eye mask (in a plastic wallet, with instructions) and will be informed about their use.

On the next morning (i.e. after the first night in hospital) the patient will be approached and asked if he or she agrees to provide outcome information. Specifically patients who were unable to give consent initially (or do not recall doing so) will have the project explained again.

Provided the patient agrees, he or she will be given a SleepSure questionnaire to answer (with help if needed); this asks about quality and quantity of sleep, and use of aids to sleep.

After discharge a researcher will also extract from the patient's clinical record (which is on computer, not paper) information such as length of stay and use of night sedation (zopiclone). Basic demographic data will be extracted, and the hospital's incident reporting system (also on computer) will be checked to identify any falls.

All data will be recorded on a computerised data-base, anonymously, and the primary analysis will be a comparison of the two groups in terms of sleep quality, with secondary analyses investigating differences in rate of recorded falls, total amount of sleep medication used during hospital stay, and length of stay

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age.
* Be expected to stay in Oxford University Hospitals National Health Service (NHS) Foundation Trust for at least one night.
* Be able to understand and use earplugs and eye mask.
* Have basic understanding of English reading and writing.
* Be considered likely to have the Mental Capacity to give consent for use of personal data in the study at the point of filling in the SleepSure Questionnaire (time of discharge). Data will not be collected from individuals who are unable to give consent with the filling in of the SleepSure questionnaire.
* Be expected to be able to fill in the SleepSure Questionnaire at the point of discharge with or without assistance.

Exclusion Criteria:

* They have or are expected to have an obvious medical contra-indication to the use of earplugs and eye mask at the point of enrollment e.g. eye infection, as per clinical judgement of recruiter.
* They are unlikely to benefit from the intervention in the judgement of the recruiter (i.e. individuals who are deaf and blind).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2016-11-25 (Actual); Primary Completion 2017-02-13 (Actual); Study Completion 2017-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derick T Wade, MD, Principal Investigator — Oxford Centre for Enablement, Oxford University Hospitals NHS FT, Windmill Road, Oxford OX3 7HE, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan is in place, but definitely data will be made available to anyone making a legitimate request

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Started 25 November 2016, Ended 13 February 2017 Recruited from medical and surgical wards in a large acute teaching and academic hospital in United Kingdom (UK)
Period: Overall Study
Arm/Group | Control | Eye Mask and Ear Plugs
Started | 97 | 109
Completed | 87 | 91
Not Completed | 10 | 18
Not completed — Discharged before night | 2 | 6
Not completed — Incomplete completion of questionnaire | 2 | 3
Not completed — No outcome; discharged or refused | 6 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Eye Mask and Ear Plugs | Total
Number analyzed (Participants) | 97 | 109 | 206
Age, Continuous [Mean (Full Range); unit: years] | 55.3 [18 to 95] | 48.4 [21 to 87] | 51.6 [18 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 70 | 121
  Male | 46 | 39 | 85
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 97 | 109 | 206
Ward type [Count of Participants; unit: Participants]
  Surgical wards | 53 | 54 | 107
  Neuroscience | 21 | 21 | 42
  Gynaecology | 14 | 26 | 40
  Acute medical | 5 | 6 | 11
  Geriatric | 4 | 2 | 6
Night after admission [Count of Participants; unit: Participants]
  First night | 6 | 4 | 10
  Second night | 41 | 52 | 93
  Third night | 9 | 16 | 25
  Fourth night | 12 | 7 | 19
  Fifth night | 8 | 6 | 14
  sixth or later night | 13 | 12 | 25
  No data returned | 6 | 9 | 15
  Discharged before first night | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: SleepSure (Questionnaire). A Short Questionnaire of the Quality and Quantity of Sleep, and Use of Aids.
Description: SleepSure is a short questionnaire which asks the patient to rate their sleep using a 1-10 numerical rating scale for eight items covering the quality of their sleep (e.g. difficulty getting to sleep, interruptions). Two additional questions recorded the use of aids. It takes no more that 2-3 minutes to complete. The eight numerical rating scores are summed and divided by 8 to give a score from 1 (very good sleep) to 10 (very poor sleep).
Time Frame: At end of first night in hospital after recruitment (i.e. the next morning)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Eye Mask and Ear Plugs
Number analyzed (Participants) | 87 | 91
units on a scale | 5.09 (2.05) | 6.33 (2.13)

2. Secondary Outcome: Length of Stay
Description: Time in days from admission to discharge from hospital (not from ward). These data were derived from the hospital administration data-base.
Time Frame: From date of admission to date of discharge, up to 90 days
Population: All patients were analysed. Two patients (one in each group) had not been discharged when data collection ended. In that instance, the number of days from recruitment to the end-of-study date was used.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control | Eye Mask and Ear Plugs
Number analyzed (Participants) | 97 | 109
days | 4.83 (6.21) | 3.67 (3.71)

3. Secondary Outcome: Use of Zopiclone (Night Sedation)
Description: The number of patients taking zopiclone during their stay. Data was taken from the Electronic patient record and was not available for any patient not discharged at the end of the study (one in each group).
  NOT the original intention of measuring "the total dose of zopiclone taken during the admission will be recorded; this is available from the electronic drug chart used in the hospital"
Time Frame: From date of admission to date of discharge, up to 90 days
Population: All patients were analysed. Two patients had not been discharged (one in each group) when data collection ended. In that instance, the number of doses of zopiclone could not be ascertained, and zero was used in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Eye Mask and Ear Plugs
Number analyzed (Participants) | 97 | 109
Participants | 2 | 3

4. Secondary Outcome: Number of Falls
Description: The number of falls, if any, will be extracted from the hospital incident recording system for the patient at the time of discharge. The data will be reported simply as the number of patients experiencing a fall; not the total number of falls experienced by the patients who had a fall. The data were taken from the electronic patient records and were not available for patients (n = 2) still in hospital at the time of discharge.
Time Frame: From date of admission to date of discharge, up to 90 days
Population: All patients were analysed. Two patients, one in each group, had not been discharged when data collection ended and data on falls were not available. The value of zero falls was used.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Eye Mask and Ear Plugs
Number analyzed (Participants) | 97 | 109
Participants | 0 | 0

5. Other Pre Specified Outcome: Use of Intervention
Description: The SleepSure questionnaire asks about use of the intervention on the night before.
Time Frame: At end of first night in hospital (first morning in hospital)
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Eye Mask and Ear Plugs
Number analyzed (Participants) | 97 | 109
Participants
  Ear plugs AND eye masks | 0 | 65
  Ear plugs ONLY | 1 | 1
  Eye mask ONLY | 1 | 13
  Neither ear plug or mask | 87 | 15
  Unknown | 8 | 15

ADVERSE EVENTS:
Time Frame: The time frame was the period of inpatient care (i.e. from the time of recruitment to the time of discharge). Two patients remained in hospital at the end of the study data collection period, and for those two patients data in the hospital incident record up to that date was used.
Description: The hospital electronic incident system records all reported incidents, which are defined as unexpected events outside normal care pathways. This would (should) record all falls, and any other adverse events. If a patient died during the admission, the 'discharge' is recorded as a death. There was no prospective study-specific data collection on each patient. No incidents (adverse events) were recorded for any patient over the course of the study.
Arm/Group | Control | Eye Mask and Ear Plugs
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/109
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/109
Other Adverse Events (participants affected / at risk) | 0/97 | 0/109

LIMITATIONS AND CAVEATS:
Less than 400 (target) recruited due to finances insufficient and delays in starting

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT02732912/Prot_SAP_000.pdf